CLINICAL TRIAL: NCT05771987
Title: Permanent Pacing as a Treatment for Drug-refractory Symptomatic Patients With Obstructive Hypertrophic Cardiomyopathy.
Brief Title: Permanent Pacing for Drug-refractory Symptomatic Patients With Obstructive Hypertrophic Cardiomyopathy.
Acronym: PACE-OHCM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09C826
Record Dates: First submitted 2023-03-06; First posted 2023-03-16 (Actual); Last update posted 2023-03-16 (Actual); Status verified 2023-03

CONDITIONS: Obstructive Hypertrophic Cardiomyopathy
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HCM patients with LVOT obstruction (Experimental): Patients with obstructive HCM are considered for this study if 1) symptomatic, 2) refractory to optimized medical therapy and 3) not or poorly* eligible for septal myectomy or with an indication to implant a pacing device (pacemaker or ICD) independent on the ventricular obstruction.
  Interventions: Procedure: pace maker implant guided by acute hemodynamic testing

INTERVENTIONS:
Procedure: pace maker implant guided by acute hemodynamic testing — To evaluate the ability of acute hemodynamic testing to optimize pacing therapy and to predict the response of HOCM to pacing

SUMMARY:
The present trial is undertaken as a pilot study on selected patients, to evaluate the ability of acute hemodynamic testing to optimize pacing therapy and to predict the response of Obstructive Hypertrophic Cardiomyopathy (OHCM) to pacing, in terms of reduction of Left Ventricular Outflow Tract (LVOT) pressure gradient and functional capacity improvement.

The Primary Objective is to demonstrate a long-term reduction in LVOT obstruction at rest and/or after Valsalva/Exercise > 30% in patients responding to acute stimulation test

ELIGIBILITY:
Inclusion Criteria:

* unequivocal diagnosis of HCM, on the basis of 2-dimensional echocardiographic demonstration of a hypertrophied (wall thickness >15 mm or > 13 mm in familial HOCM) and non dilated LV in the absence of another cardiac or systemic disease capable of producing the same magnitude of hypertrophy;
* patients in whom coronary disease has been excluded;
* presence of severe refractory symptoms (NYHA class II-IV), as evidenced by moderate-to-severe functional disability resulting from exertional dyspnea or chest pain sufficient to support a desire for alternative treatment modalities, following administration (in standard dosages) of beta-blocker and either disopyramide or verapamil, independently or in association;
* peak instantaneous LV outflow tract gradient > 50 mm Hg (resting or provoked), estimated by continuous wave Doppler;

Exclusion Criteria:

* end-stage phase of HCM (unless CRT therapy is considered);
* ejection fraction <50% (unless CRT therapy is considered);
* severe mitral valve disease (+++) not related to systolic anterior movement and/or papillary muscle abnormalities;
* age below 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-06-28 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Reduction of LVOT pressure gradient | 3 months
  Long-term reduction in LVOT obstruction at rest and/or after Valsalva/Exercise > 30% in patients responding to acute stimulation test

SECONDARY OUTCOMES:
Clinical improvement: change in NYHA class | 6-12 months
  Improvement of NYHA class
Clinical improvement: change in exercise capacity | 6-12 months
  6-minutes walking test
Clinical improvement: change in peak VO2 | 6-12 months
  Improvement in peak VO2
Clinical improvement: change in NT-proBNP concentration | 6-12 months
  Reduction in NT-proBNP concentration

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Auxologico Italiano, Milan, Italy

IPD SHARING:
Plan to Share IPD: No